CLINICAL TRIAL: NCT02787200
Title: Identification of Time-invariant EEG Signals for Brain-Computer Interface
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 201604024RIND
Record Dates: First submitted 2016-05-26; First posted 2016-06-01 (Estimated); Last update posted 2016-06-08 (Estimated); Status verified 2016-06

CONDITIONS: EEG Data Analysis; Healthy Subjects
Keywords: electroencephalogram (EEG),Human brain,Brain-Computer Interface

STUDY DESIGN:
Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

SUMMARY:
This study aims to identify various time-variant and time-invariant components of EEG signals using advanced signal processing techniques, such as machine learning. The investigators' ultimate goal is to develop universal or customised brain-computer interface that are stable across days or even years.

ELIGIBILITY:
Exclusion criteria:

1. Severe vision disorders which prevent volunteers to recognize instructions on the screen
2. Severe psychiatric disorders
3. Severe sleep disorders which keep volunteers awake for two hours
4. Volunteers with claustrophobia
5. Patients who underwent stroke and brain surgery
6. Patients with neuromuscular diseases

Ages: 20 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Healthy volunteers that understands Mandarin instructions.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2016-05; Primary Completion 2017-05 (Estimated); Study Completion 2017-05 (Estimated)

PRIMARY OUTCOMES:
Time invariant components of EEG signals | One month

CONTACTS AND LOCATIONS:
Overall Officials: Tsung-Ren Huang, Principal Investigator — National Taiwan University
Locations (1):
- National Taiwan University Hospital, Taipei, Taipei, Taiwan